CLINICAL TRIAL: NCT00103389
Title: A Phase II Study of Docetaxel With PI-88 in Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: Docetaxel With or Without PI-88 in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROGEN-PR88202; CDR0000409568 (Registry Identifier: PDQ (Physician Data Query)); AUS-RNSH-0309-183M
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — phosphomannopentaose sulfate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- docetaxel (Active Comparator): treated with docetaxel alone
  Interventions: Drug: docetaxel
- PI-88+docetaxel (Experimental): treated with docetaxel and PI-88
  Interventions: Drug: PI-88; Drug: docetaxel

INTERVENTIONS:
Drug: PI-88 — PI-88+docetaxel
  Arms: PI-88+docetaxel
Drug: docetaxel — docetaxel only

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. PI-88 may stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. It may also help docetaxel work better by making tumor cells more sensitive to the drug. Giving docetaxel together with PI-88 may kill more tumor cells. It is not yet known whether giving docetaxel together with PI-88 is more effective than docetaxel alone in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying docetaxel and PI-88 to see how well they work when given together compared to docetaxel alone in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety and efficacy of docetaxel with vs without PI-88 in patients with stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the efficacy markers of docetaxel and PI-88 in these patients.
* Determine the safety and potential efficacy of PI-88 alone as maintenance therapy in patients whose disease has been controlled with docetaxel and PI-88 combination therapy.
* Determine the safety and potential efficacy of PI-88 alone as third-line therapy in these patients.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on days 1, 8, and 15.
* Arm II: Patients receive docetaxel as in arm I. Patients also receive PI-88 subcutaneously once daily on days 1-4, 8-11, and 15-18.

In both arms, treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients in arm II with stable or responding disease after 6 courses may continue to receive PI-88 alone as maintenance therapy. Patients in arm I with progressive disease or unacceptable toxicity before the completion of 6 courses may receive PI-88 alone as third-line therapy.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Stage IIIB or IV disease
* Eligible for second-line docetaxel

  * Disease progression during or after completion of prior first-line therapy comprising radiotherapy and/or platinum-based chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 2 months

Hematopoietic

* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* No history of thrombotic thrombocytopenic purpura or other platelet disease

Hepatic

* Bilirubin normal
* ALT and AST ≤ 2.5 times upper limit of normal (ULN) (1.5 times ULN if alkaline phosphatase > 2.5 times ULN)
* Alkaline phosphatase ≤ 5 times ULN (unless bone metastases are present)
* PT < 1.5 times ULN
* Activated PTT normal

Renal

* Creatinine clearance or glomerular filtration rate > 50mL/min

Cardiovascular

* None of the following within the past 3 months:

  * Myocardial infarction
  * Stroke
  * Congestive heart failure

Immunologic

* No history of immune-mediated thrombocytopenia
* No evidence of anti-heparin antibodies
* No history of allergy and/or hypersensitivity to anti-coagulants or thrombolytic agents, especially heparin
* No history of allergy to polysorbate 80
* No uncontrolled or serious infection within the past 4 weeks

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior docetaxel

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior radiotherapy to > 30% of marrow-bearing bone
* Concurrent local palliative radiotherapy allowed

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 4 weeks since prior antineoplastic therapy
* More than 2 weeks since prior and no concurrent heparin or low-molecular weight heparin
* More than 4 weeks since prior investigational therapy
* No concurrent aspirin or aspirin-containing medications except low-dose aspirin (≤ 100 mg/day)
* No concurrent nonsteroidal anti-inflammatory drugs except cyclooxygenase-2 inhibitors
* No concurrent warfarin or warfarin-containing medications except low-dose warfarin (≤ 1 mg/day)
* No concurrent antiplatelet drugs, including any of the following:

  * Abciximab
  * Clopidogrel
  * Dipyridamole
  * Ticlopidine
  * Tirofiban
* No concurrent drugs that may inhibit docetaxel metabolism, including any of the following:

  * Cyclosporine
  * Terfenadine
  * Ketoconazole
  * Erythromycin
  * Troleandomycin
* No other concurrent investigational drugs
* No other concurrent antineoplastic therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are progression-free as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v2.0 at 6 months
Non-progression rate as measured by RECIST v2.0 at 6 months

SECONDARY OUTCOMES:
Time to progression as measured by RECIST v2.0 at baseline, and then week 4 of courses 2, 3, 4, and 6
Response rate as measured by RECIST v2.0 at baseline, and then week 4 of courses 2, 3, 4, and 6
Quality of life as measured by Lung Cancer Symptom Scale (LCSS) every month
Overall survival as measured by RECIST v2.0 at death

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, MD, Study Chair — Royal North Shore Hospital
Locations (13):
- Australia (13):
  - Sydney Heamatology and Oncology Clinics, Hornsby, New South Wales
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Mater Medical Centre, South Brisbane, Queensland
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Murray Valley Private Hospital and Cancer Treatment Centre, Wodonga, Victoria
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No